CLINICAL TRIAL: NCT07381023
Title: Effectiveness of Heart Rate Variability in Reducing Anxiety in Pre-Heart Transplant Candidates in the ICU
Brief Title: Using Breathing Techniques to Ease Anxiety in ICU Patients Awaiting Heart Transplants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford HealthCare (Other)
Responsible Party: Principal Investigator, Rachel Cavallaro, Principal Investigator, Hartford HealthCare
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HHC-2025-0188
Record Dates: First submitted 2025-10-01; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Anxiety; Heart Transplant Patients
Keywords: Heart Transplant Candidates; Heart Rate Variability Biofeedback; Anxiety; Breathing techniques; Behavioral Health in Transplant; Cardiac Anxiety; Biofeedback Therapy
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heart Rate Variability Biofeedback for Anxiety Reduction in ICU Heart Transplant Candidates" (Experimental): Participants in this arm will receive a single-session heart rate variability biofeedback (HRVB) intervention while admitted to the intensive care unit (ICU) as candidates for heart transplantation. The intervention includes a guided breathing exercise using a biofeedback device or app that provides real-time feedback on heart rate and breathing patterns. A trained clinician will lead the session, which is designed to promote autonomic regulation and reduce anxiety. Participants will complete self-report anxiety assessments immediately before and after the session to evaluate changes in psychological distress. They will also receive brief instruction on how to continue using the breathing technique independently as appropriate.
  Interventions: Behavioral: Heart Rate Variability Biofeedback (HRVB)

INTERVENTIONS:
Behavioral: Heart Rate Variability Biofeedback (HRVB) — Participants will receive a single-session heart rate variability biofeedback (HRVB) intervention while admitted to the intensive care unit (ICU) as candidates for heart transplantation. The intervention involves guided paced breathing using a biofeedback device or app that provides real-time feedback on heart rate and breathing patterns. A trained clinician will lead the session, which is designed to promote autonomic regulation and reduce anxiety. Participants will complete pre- and post-intervention self-report assessments to evaluate changes in anxiety levels. They will also receive brief instruction on how to continue using the breathing technique independently.

SUMMARY:
The goal of this clinical trial is to learn whether a breathing-based relaxation technique called heart rate variability biofeedback (HRVB) can help reduce anxiety in adult patients who are in the intensive care unit (ICU) and waiting for a heart transplant. The main questions it aims to answer are:

Can HRVB reduce anxiety in patients awaiting heart transplantation in the ICU? Does HRVB help patients feel more in control of their emotions during this stressful time?

Participants will:

Complete a brief anxiety assessment before and after the intervention Participate in a guided HRVB session using a breathing device or app Learn how to use the technique on their own for future stress management

DETAILED DESCRIPTION:
This is a single-group clinical trial designed to evaluate the effectiveness of heart rate variability biofeedback (HRVB) in reducing anxiety among adult patients who are currently admitted to the intensive care unit (ICU) and awaiting heart transplantation. Patients in this population often experience elevated levels of psychological distress, including anxiety and panic symptoms, due to the uncertainty of their medical condition, the high-stress ICU environment, and the emotional burden of awaiting a life-saving procedure.

Heart rate variability (HRV) is a physiological marker of autonomic nervous system function and emotional regulation. HRVB is a non-invasive intervention that teaches individuals to regulate their breathing in a way that promotes optimal HRV. This technique has been shown in prior research to reduce anxiety and improve emotional resilience in various populations, but its application in critically ill transplant candidates remains underexplored.

Participants in this study will complete a baseline assessment of anxiety using validated self-report measures. They will then participate in a guided HRVB session, which includes paced breathing instruction and the use of a biofeedback device or app that provides real-time feedback on heart rate and breathing patterns. Following the session, participants will complete a post-intervention assessment to evaluate changes in anxiety levels. Participants will also be encouraged to continue practicing the technique independently as appropriate.

The primary outcome is the change in self-reported anxiety from pre- to post-intervention. Secondary outcomes may include changes in perceived emotional control and physiological indicators of stress. This study aims to assess the feasibility and immediate psychological benefits of HRVB in a high-acuity medical setting and to inform future research on integrative behavioral health interventions for transplant candidates.

ELIGIBILITY:
Inclusion Criteria

* any gender
* any race/ethnicity
* ≥18 years old with no upper limit
* currently inpatient in the cardiac ICU, awaiting heart transplant
* elevated anxiety symptoms as evidenced by cut scores on the Depression, Anxiety and Stress Scale (DASS-21) and the Cardiac Anxiety Questionnaire (CAQ) (Lovibond & Lovibond, 1995; Eifert et al., 2000).
* proficiency in speaking, reading and writing in English Participants in this study must be proficient in English due to the language limitations of the study administrator. The intervention includes a teaching component that requires verbal instruction, psychoeducation, and interactive engagement, all of which will be conducted exclusively in English. At this time, the study administrator is only proficient in English and is unable to reliably deliver the intervention or assess participant understanding in other languages. To ensure consistency, accuracy, and fidelity of the intervention, as well as to maintain ethical standards in informed consent and participant comprehension, only English-speaking individuals will be eligible to participate.
* able/willing to consent to participate Exclusion Criteria
* <18 years of age
* active psychosis or delirium
* current neurological problems (e.g., stroke) at time of enrollment that would interfere with the ability to complete the practice
* on a ventilator at time of enrollment
* pregnancy
* unable or unwilling to consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
DASS-21 Anxiety Scale | Baseline (pre-intervention) and after 2 weeks (post-intervention)
  Standardized self-report measure of anxiety

SECONDARY OUTCOMES:
Cardiac Anxiety Questionnaire | Baseline (pre-intervention) and after 2 weeks (post-intervention)
  Standardized self-report measure of anxiety

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 1 year after publication with no end date